CLINICAL TRIAL: NCT05780541
Title: A Multicenter, Adaptive, Randomized, Blinded Controlled Trial of the Safety and Efficacy of Investigational Therapeutics for Hospitalized Patients With COVID-19 (Trial H6: PF-07304814)
Brief Title: PF-07304814 for Inpatients With COVID-19 (An ACTIV-3/TICO Treatment Trial)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The agent was withdrawn from development by the manufacturer after being placed on clinical hold by the US FDA.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: International Network for Strategic Initiatives in Global HIV Trials (INSIGHT) (Network); University of Copenhagen (Other); Medical Research Council (Other Government); Kirby Institute (Other Government); Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency); Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network); National Heart, Lung, and Blood Institute (NHLBI) (NIH); US Department of Veterans Affairs (U.S. Federal Agency); Prevention and Early Treatment of Acute Lung Injury (Other); Cardiothoracic Surgical Trials Network (Other); Pfizer (Industry); University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 014/ACTIV-3/H6
Record Dates: First submitted 2023-03-20; First posted 2023-03-22 (Actual); Results first posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: COVID-19
Keywords: COVID-19; COVID 19; Coronaviridae Infections; Coronavirus Infections; RNA Virus Infections; Virus Diseases; Nidovirales Infections; SARS-CoV-2; SARS Coronavirus; ACTIV-3; ACTIV3; TICO
MeSH Terms: conditions — COVID-19; Coronaviridae Infections; Coronavirus Infections; RNA Virus Infections; Virus Diseases; Nidovirales Infections; Severe Acute Respiratory Syndrome | interventions — lufotrelvir; remdesivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PF-07304814 plus SOC (Experimental): * PF-07304814 250 mg per day for 5 days; administered as a constant rate IV infusion
  * Remdesivir is provided to all study participants as SOC unless contraindicated for an individual patient; administered by IV infusion
  Interventions: Drug: PF-07304814; Biological: Remdesivir
- Placebo plus SOC (Placebo Comparator): * Placebo administered by IV infusion
  * Remdesivir is provided to all study participants as SOC unless contraindicated for an individual patient; administered by IV infusion
  Interventions: Drug: Placebo; Biological: Remdesivir

INTERVENTIONS:
Drug: PF-07304814 — PF-07304814 is a phosphate ester prodrug of PF-00835231 (active moiety), a potent and selective inhibitor of the SARS-CoV-2 3CLpro.
  Arms: PF-07304814 plus SOC
Drug: Placebo — Commercially available 0.9% sodium chloride solution
  Arms: Placebo plus SOC
Biological: Remdesivir — Antiviral agent
  Other Names: Veklury

SUMMARY:
This study looks at the safety and effectiveness of PF-07304814 in treating COVID-19 in people who have been hospitalized with the infection. Participants in the study will be treated with either PF-07304814 plus current standard of care (SOC), or with placebo plus current SOC. This is ACTIV-3/TICO Treatment Trial H6.

DETAILED DESCRIPTION:
This is a treatment trial of the ACTIV-3/TICO master protocol (NCT04501978) to evaluate the safety and efficacy of PF-07304814 in hospitalized patients infected with COVID-19.

This is a randomized, blinded, controlled sub-study of PF-07304814 plus current SOC against placebo plus current SOC. The placebo arm may be shared across other sub-studies of the ACTIV-3/TICO master protocol. When more than one drug is being tested at the same time, participants will be randomly allocated to treatments or placebo.

Randomization will be stratified by study site pharmacy and disease severity. There are 2 disease severity strata: participants without organ failure (severity stratum 1) and participants with organ failure (severity stratum 2).

An independent Data and Safety Monitoring Board (DSMB) will regularly review interim analyses and summarize safety and efficacy outcomes. The pace of enrollment with be initially restricted, and there will be an early review of safety data by the DSMB. At the outset of the trial, only participants in disease severity stratum 1 will be enrolled. This will continue until approximately 300 participants are enrolled and followed for 5 days. The exact number will vary according to the speed of enrollment and the timing of DSMB meetings. Prior to expanding enrollment to also include patients in disease severity stratum 2, safety will be evaluated and a pre-specified futility assessment by the DSMB will be carried out using 2 ordinal outcomes assessed at Day 5.

If PF-07304814 passes the futility assessment, enrollment of participants will be expanded, seamlessly and without any data unblinding, to include participants in disease severity stratum 2 as well as those in disease severity stratum 1. Future interim analyses will be based on the primary endpoint of sustained recovery and will use pre-specified guidelines to determine early evidence of benefit, harm, or futility for the investigational agent. Participants will be followed for 18 months following randomization.

This trial will be conducted in several hundred clinical sites. Participating sites are affiliated with networks funded by the United States National Institutes of Health (NIH) and the US Department of Veterans Affairs.

ELIGIBILITY:
Inclusion Criteria: Refer to the master protocol (NCT04501978)

Exclusion Criteria: Refer to the master protocol (NCT04501978)

Additional Exclusion Criteria:

1. Participants with moderate to severe hepatic impairment (i.e. Child-Pugh class B or C) or acute liver failure.
2. Participants receiving any medications or substances that are strong inhibitors or inducers of cytochrome P450 (CYP) 3A4 (see Section H6.3.4).
3. Patients will be excluded if taking drugs which have a narrow therapeutic window that are substrates of CYP3A4, including but not limited to: astemizole, cisapride, cyclosporine, dihydroergotamine, ergotamine, pimozide, quinidine, sirolimus, tacrolimus, and terfenadine.
4. Pregnant women
5. Nursing mothers
6. Women of child-bearing potential who are unwilling to acknowledge the strong advice to abstain from sexual intercourse with men or practice appropriate contraception through 5 weeks of the study.
7. Men who are unwilling to acknowledge the strong advice to abstain from sexual intercourse with women of child-bearing potential or to use barrier contraception through 5 weeks of the study.
8. Patients with a history of deep vein thrombosis or pulmonary thrombotic embolism*.

   * Prior to the initial futility assessment, which is performed when approximately 150 patients have been enrolled on PF-07304814 and 150 on placebo, patients with a history of deep vein thrombosis or pulmonary embolism will be excluded. These patients will be eligible for the trial if the initial futility assessment is passed by this agent, and if risk-benefit is favorable based on an assessment of available data that is reviewed by the independent DSMB. These data will include treatment comparisons of thromboembolic events and coagulation markers, and any additional data from studies carried out by Pfizer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2023-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Lundgren, Prof., Principal Investigator — INSIGHT Copenhagen International Coordinating Centre, Rigshospitalet, University of Copenhagen; James Neaton, Prof., Study Chair — INSIGHT Statistical and Data Management Center, University of Minnesota
Locations (40):
- United States (31):
  - Velocity Chula Vista (Site 080-034), 752 Medical Center Ct., Ste. 304, Chula Vista, California
  - Cedars-Sinai Medical Center (Site 208-002), 8700 Beverly Blvd., Los Angeles, California
  - Sacramento VA Medical Center (Site 074-023), 10535 Hospital Way, Mather, California
  - Hoag Memorial Hospital Presbyterian (Site 080-026), One Hoag Drive, Newport Beach, California
  - Palo Alto VAMC (Site 074-005), 3801 Miranda Avenue, Palo Alto, California
  - UC Davis Health (Site 203-004), 2315 Stockton Blvd., Sacramento, California
  - VA San Diego Healthcare System (Site 074-016), 3350 La Jolla Village Drive, San Diego, California
  - San Francisco VAMC (Site 074-002), 4150 Clement St., San Francisco, California
  - National Jewish Health / St. Joseph Hospital (Site 204-003), 1400 Jackson Street, Denver, Colorado
  - West Haven VA Medical Center (Site 025-007), 950 Campbell Avenue, West Haven, Connecticut
  - MedStar Health Research Institute (Site 009-021), MedStar Washington Hospital Center, 110 Irving St., NW., Washington D.C., District of Columbia
  - Bay Pines VAMC (Site 074-004), 10000 Bay Pines Blvd., Bldg. 100, Room 5B-104, Bay Pines, Florida
  - Hillsborough County Health Department, University of South Florida (Site 032-001), Tampa, Florida
  - Lutheran Medical Group (Site 301-010), 7916 W. Jefferson Boulevard, Fort Wayne, Indiana
  - Ochsner Clinic Foundation (Site 301-015), 1514 Jefferson Highway, New Orleans, Louisiana
  - Massachusetts General Hospital (Site 202-002), 55 Fruit Street, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center (Site 202-001), 330 Brookline Ave., Boston, Massachusetts
  - Henry Ford Health System, Henry Ford Hospital (Site 014-001), 2799 W. Grand Blvd., Detroit, Michigan
  - Dartmouth-Hitchcock Medical Center/Mary Hitchcock Memorial Hospital (Site 301-024), One Medical Center Drive, Lebanon, New Hampshire
  - Duke University Hospital (Site 301-006), 2301 Erwin Road, Durham, North Carolina
  - Portland VA Healthcare System (Site 074-024), 3710 SW. US Veterans Hospital Road, Portland, Oregon
  - Rhode Island Hospital (Site 080-036), 593 Eddy Street, Providence, Rhode Island
  - The Miriam Hospital (Site 080-039), 164 Summit Ave., Providence, Rhode Island
  - Ralph H. Johnson VA Medical Center (Site 074-015), 109 Bee Street, Charleston, South Carolina
  - MUSC Research Nexus Clinic (Site 210-002), 96 Jonathan Lucas St., CSB 214, Charleston, South Carolina
  - MUSC Health Florence Medical Center (Site 210-006), 805 Pamplico Highway, Florence, South Carolina
  - Parkland Health and Hospital Systems (Site 084-002), 5200 Harry Hines Blvd, Dallas, Texas
  - UT Southwestern Medical Center (Site 084-001), 1936 Amelia Court, 2nd Floor, Dallas, Texas
  - Baylor, Scott and White Health (Site 301-003), Baylor University Medical Center, 3500 Gaston Ave., Dallas, Texas
  - University of Utah Hospital (Site 211-002), 419 Wakara Way, Suite 207, Salt Lake City, Utah
  - West Virginia University (Site 301-023), One Medical Center Drive, Morgantown, West Virginia
- Denmark (9):
  - Aalborg Hospital (Site 625-005), Hobrovej 18, Aalborg
  - Aarhus Universitetshospital, Skejby (Site 625-002), Department of Infectious Diseases, Palle Juul-Hensens Boulevard 99, Aarhus N
  - Bispebjerg Hospital (Site 625-013), Bispebjerg Bakke 23, Copenhagen
  - Righospitalet (Site 625-006), Blegdamsvej 9,, Copenhagen Ø
  - Herlev/Gentofte Hospital (Site 625-012), Medicinsk Afdeling, Herlev Ringvej 75, Herlev
  - Nordsjællands Hospital (Site 625-009), Dyrehavevej 29, Hillerød
  - Kolding Sygehus (Site 625-011), Medicinsk Afdeling, Sygehusvej 24, Kolding
  - Odense University Hospital (Site 625-004), Infektionsmedicinsk Forskningsenhed, J.B. Winsløwsgade 4, Odense
  - Zealand University Hospital, Roskilde (Site 625-010), Sygehusvej 10, Roskilde

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 40 sites in 2 countries (Denmark, USA). The first subject was enrolled on 15 Sep 2021 and the last subject was enrolled on 29 Dec 2021.
Pre-assignment Details: Of 58 subjects enrolled, 58 met inclusion criteria and were randomized to treatment.
Groups:
- PF-07304814 Plus SOC: * PF-07304814 250 mg per day for 5 days; administered as a constant rate IV infusion
  * Remdesivir is provided to all study participants as SOC unless contraindicated for an individual patient; administered by IV infusion
  PF-07304814: PF-07304814 is a phosphate ester prodrug of PF-00835231 (active moiety), a potent and selective inhibitor of the SARS-CoV-2 3CLpro.
  Remdesivir: Antiviral agent
- Placebo Plus SOC: * Placebo administered by IV infusion
  * Remdesivir is provided to all study participants as SOC unless contraindicated for an individual patient; administered by IV infusion
  Placebo: Commercially available 0.9% sodium chloride solution
  Remdesivir: Antiviral agent
Period: Overall Study
Arm/Group | PF-07304814 Plus SOC | Placebo Plus SOC
Started | 32 | 26
Completed | 32 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-07304814 Plus SOC | Placebo Plus SOC | Total
Number analyzed (Participants) | 32 | 26 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (13.2) | 59.5 (16.6) | 60.3 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 14 | 23
  Male | 23 | 12 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 8 | 20
  Not Hispanic or Latino | 20 | 18 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 20 | 19 | 39
  More than one race | 0 | 0 | 0
  Other | 2 | 0 | 2
  Only ethnicity reported | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sustained Recovery
Description: Sustained recovery defined as being discharged from the index hospitalization, followed by being alive and home for 14 consecutive days prior to Day 90.
Time Frame: Through Day 90
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07304814 Plus SOC | Placebo Plus SOC
Number analyzed (Participants) | 32 | 26
Participants | 23 | 13

2. Primary Outcome: Number of Participants With an Ordinal Outcome on Day 5
Description: Ordinal outcome with 7 mutually exclusive categories
Time Frame: Status on Day 5
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07304814 Plus SOC | Placebo Plus SOC
Number analyzed (Participants) | 32 | 26
Participants
  7 = Death | 0 | 4
  6 = Invasive ventilation, ECMO, mechanical circulatory support, new renal replacement therapy | 5 | 3
  5 = Non-invasive ventilation or high flow oxygen | 11 | 5
  4 = Supplement oxygen (≥4 L/min or ≥4 L/min above baseline, but not high flow oxygen) | 5 | 5
  3 = Supplement oxygen (<4 L/min or <4 L/min above baseline, but not high flow oxygen) | 5 | 0
  2 = Limiting symptoms due to COVID-19, but no need of new or increased oxygen from baseline | 3 | 4
  1 = No limiting symptoms due to COVID-19 | 3 | 5

3. Secondary Outcome: Number of Participants Who Died From All Causes
Description: All-cause mortality
Time Frame: Through Day 90
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07304814 Plus SOC | Placebo Plus SOC
Number analyzed (Participants) | 32 | 26
Participants | 9 | 6

4. Secondary Outcome: Number of Participants With a Safety Outcome Through Day 5
Description: Death, SAE, clinical organ failure, serious infections, or Grade 3 or 4 event through Day 5
Time Frame: Through Day 5
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07304814 Plus SOC | Placebo Plus SOC
Number analyzed (Participants) | 32 | 26
Participants | 12 | 10

5. Secondary Outcome: Number of Participants With a Safety Outcome Through Day 28
Description: Death, SAE, clinical organ failure, serious infections, or Grade 3 or 4 event through Day 28
Time Frame: Through Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07304814 Plus SOC | Placebo Plus SOC
Number analyzed (Participants) | 32 | 26
Participants | 17 | 11

6. Secondary Outcome: Number of Participants With a Safety Outcome Through Day 90
Description: Death, SAE, clinical organ failure, serious infections through Day 90
Time Frame: Through Day 90
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07304814 Plus SOC | Placebo Plus SOC
Number analyzed (Participants) | 32 | 26
Participants | 15 | 11

ADVERSE EVENTS:
Time Frame: 90 Days
Description: Only Grade 3 or 4 AEs were collected.
Arm/Group | PF-07304814 Plus SOC | Placebo Plus SOC
All-Cause Mortality (participants affected / at risk) | 9/32 | 6/26
Serious Adverse Events (participants affected / at risk) | 2/32 | 1/26
Other Adverse Events (participants affected / at risk) | 11/32 | 9/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PF-07304814 Plus SOC (N=32) | Placebo Plus SOC (N=26)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PF-07304814 Plus SOC (N=32) | Placebo Plus SOC (N=26)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal hematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (1)
Oedema (General disorders) | 0 (0) | 1 (2)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 2 (2)
Labile blood pressure (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol: Trial H6 Protocol (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT05780541/Prot_000.pdf
  • Study Protocol: Master Protocol (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT05780541/Prot_001.pdf
  • Statistical Analysis Plan (2022-02-23): https://cdn.clinicaltrials.gov/large-docs/41/NCT05780541/SAP_002.pdf
  • Informed Consent Form (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT05780541/ICF_003.pdf